CLINICAL TRIAL: NCT02871180
Title: A Late Night Snack May be Necessary to Prevent Nocturnal Hyperglycemia in Type 1-diabetic Patients Using Insulin Glargine (LANTUS)
Brief Title: Late Night Snack and Insulin Glargine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabeteszentrum Bad Lauterberg im Harz (Other)
Responsible Party: Principal Investigator, Michael A. Nauck, Prof. Dr. med. Michael A. Nauck, Diabeteszentrum Bad Lauterberg im Harz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Late night snack & Lantus
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: Hypoglycemia; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With late night snack (Other): At 10 p.m. a late night snack (one slice of whole meal rye bread containing approximately 20 g of carbohydrate) was eaten from Type 1 diabetic patients on an intensified conventional treatment regimen.
  Interventions: Dietary Supplement: Late night snack
- Without late night snack (Other): Not nutrients (No late night snack) were consumed at 10 p.m. from Type 1 diabetic patients on an intensified conventional treatment regimen..
  Interventions: Other: No late night snack

INTERVENTIONS:
Dietary Supplement: Late night snack — The late night snack was one slice of whole meal rye bread containing approximately 20 g of carbohydrate.
  Arms: With late night snack
Other: No late night snack — Patient consumed no nutrients at late night.
  Arms: Without late night snack

SUMMARY:
Twenty patient with Type 1 diabetes, using insulin glargine as basal insulin, participated in a prospective, controlled crossover trial comparing blood glucose profiles over two 24 h periods with and without a late night snack (a slice of rye bread, 20 g carbohydrates, at 10 p.m.), in randomized order. The main endpoint was the number of hypoglycemic episodes with a confirmed laboratory blood glucose ≤ 50 mg/dl between 10 p.m. and 8 p.m. the following day. Secondary endpoint was the blood glucose profile during this period.

DETAILED DESCRIPTION:
The order of studies (with and without a late night snack) was determined by randomization. Study-related procedures started at 6 p.m. (standard blood glucose profiles with determinations at 6, 8, and 10 p.m, at midnight, at 2, 4, 6:45, 8:45 a.m., and at noon and 2, 6, and 8 p.m. of the following day). At 10 p.m. a late night snack (one slice of whole meal rye bread containing approximately 20 g of carbohydrate) was eaten or no nutrients were consumed, as determined by the randomization protocol. After one day without study-related activities, the study was repeated with the complementary protocol (crossover design). Patients were instructed to use fast-acting insulin to correct hyperglycemia three times per day (before major meals) or to take in additional carbohydrate when symptomatic or chemical hypoglycemia was noted. They were asked not to perform strenuous exercise beyond their normal daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Basal insulin substitution with insulin glargine at least 3 month

Exclusion Criteria:

* Severe disorders
* Severe and clinical significant gastroparesis
* History of pancreatitis or pancreatic cancer
* Severe Liver disorder (liver enzymes > three times upper normal limit)
* Pregnancy
* Drug- or alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-03; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia | 26 hours
  Hypoglycemia with a plasma glucose ≤ 50 mg/dl as determined with a standardized laboratory method

SECONDARY OUTCOMES:
Blood glucose profile | 26 hours
  The blood glucose profile with and without a late-night snack . (standard blood glucose profiles with determinations at 6, 8, and 10 p.m, at midnight, at 2, 4, 6:45, 8:45 a.m., and at noon and 2, 6, and 8 p.m. of the following day).

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Nauck, Prof., Principal Investigator — St. Josef-Hospital
Locations (1):
- Diabeteszentrum Bad Lauterberg, Bad Lauterberg im Harz, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No